CLINICAL TRIAL: NCT04042974
Title: Vaginal Dinoprostone Prior to Diagnostic Office Hysteroscopy in Primarily Infertile Patients:a Randomized Controlled Trial
Brief Title: Vaginal Dinoprostone Prior to Diagnostic Office Hysteroscopy in Primarily Infertile Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dinoprostone hysteroscopy
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Hysteroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dinoprostone (Experimental): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Interventions: Drug: vaginal dinoprostone
- placebo (Placebo Comparator): one tablet of placebo inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vaginal dinoprostone — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Arms: dinoprostone
Drug: placebo — one tablet of placebo inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Arms: placebo

SUMMARY:
To compare the effectiveness of vaginal dinoprostone with placebo in minimizing the pain experienced by primarily infertile patients during diagnostic ofﬁce hysteroscopy and to assess the ease of insertion of hysteroscope as reported by the hysteroscopist.

DETAILED DESCRIPTION:
hysteroscopy is commonly used in the diagnosis and treatment of intrauterine lesions such as polyps, ﬁbroids, septa, and adhesions, and in the presence of abnormal bleeding and during the removal of an intrauterine device or foreign body. Cervical ripening is made possible by the use of medication through different routes. The most commonly used agent is misoprostol, a synthetic prostaglandin E1 (PGE1) analog that is frequently administered in off-label use in obstetrics and gynecology for medical abortion, labor induction, endometrial biopsy, dilatation and curettage, intrauterine device insertion, myomectomy, postpartum haemorrhage, and cervical ripening. In contrast, dinoprostone, a natural PGE2, is mostly used in obstetrics for cervical ripening and the stimulation of uterine contractions to induce labor.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women with primary infertility requiring a diagnostic hysteroscopy as a part of an infertility diagnosis workup

Exclusion Criteria:

* • women with suspected pregnancy

  * heavy vaginal bleeding
  * recent pelvic infection
  * those known to have hypersensitivity or contraindication to dinoprostone
  * those who received analgesics prior to OH
  * a concomitant neurologic disease that could affect the correct evaluation of pain

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-10 (Estimated); Primary Completion 2019-11-10 (Estimated); Study Completion 2019-11-20 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | an expected average of 10 minutes
  Pain intensity will be assessed by visual analogue scale during the procedure.visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Intensity of pain | 30 minutes after the procedure
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure.visual analogue scale ranging from 0 to 10
Operative time | an expected average 10 minutes
  From the introduction of hysteroscope into the vagina till compilation of hysteroscopic examination

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University